CLINICAL TRIAL: NCT01879462
Title: A Randomized, Single-Blind, Dose Escalation, First Time in Human Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Doses of GSK2878175 in Healthy Adults
Brief Title: A First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single & Repeat Escalating Doses of GSK2878175 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 116973
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C (CHC); Hepatitis C virus (HCV); NS5B; pharmacokinetics; GSK2878175; safety; FTIH; healthy subjects
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — GSK2878175

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort A (Experimental): Subjects in this cohort will receive 3 treatments (either active drug or placebo for each dose level) in 3 treatment periods (one per period). Subjects will receive GSK2878175 5 mg, GSK2878175 50 mg, and GSK2878175 200 mg in treatment period 1, 2, and 3 respectively in fasted state (with 1:3 ratio of placebo to active treatment at each treatment period).
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort B (Experimental): Subjects in this cohort will receive 3 treatments (either active drug or placebo for each dose level) in 3 treatment periods (one per period). Subjects will receive GSK2878175 15 mg in fasted state, GSK2878175 100 mg in fasted state, and GSK2878175 100 mg in fed state in treatment period 1, 2, and 3 respectively (with 1:3 ratio of placebo to active treatment at each treatment period).
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort C (Experimental): Subjects in this cohort will receive GSK2878175 15 mg single dose or placebo for 7 days in fasted state (with 1:4 ratio of placebo to active treatment).
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort D (Experimental): Subjects in this cohort will receive placebo and GSK2878175 50 mg single dose or placebo for 7 days in fasted state, (with 1:4 ratio of placebo to active treatment).
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort E (Experimental): Subjects in this cohort will receive placebo and GSK2878175 100 mg single dose or placebo for 7 days in fasted state, (with 1:4 ratio of placebo to active treatment).
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort F (Experimental): Subjects in this cohort will receive placebo and GSK2878175 200 mg single dose or placebo for 7 days in fasted state, (with 1:4 ratio of placebo to active treatment).
  Interventions: Drug: GSK2878175; Drug: Placebo

INTERVENTIONS:
Drug: GSK2878175 — Round tablets (5.0mg) given once daily single and repeated (to 7 days), Oral dose.
Drug: Placebo — Visually matching GSK2878175

SUMMARY:
GSK2878175 is a site IV NS5B non-nucleoside inhibitor (NNI) being developed for the treatment of chronic HCV infection. This study represents the first administration of GSK2878175 in humans to define safety, tolerability, and pharmacokinetics (PK) following single and repeat doses of GSK2878175 in healthy subjects.

This is a Phase 1, randomized, single-blind, placebo-controlled, dose escalation study to determine the safety, tolerability, and PK profile of GSK2878175 in single (Part 1) and repeat doses (Part 2) in healthy subjects. In addition the study will explore the effect of a moderate (30%) fat meal on single dose PK endpoints in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECGs. There should be no evidence of cardiac, pulmonary, hepatic, biliary, gastrointestinal, or renal disorders, or cancer within the past 5 years (except localized or in situ cancer of the skin). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria and are reported as outside of the normal reference range for healthy volunteers may be included only if the Investigator considers the finding is unlikely to introduce additional risk to the subject and will not interfere with the study procedures.
* Body weight >50 Kilograms(kg) (110 pounds) for men and >45kg (99pounds) women and a body mass index (BMI) between 18.5-32 kg/meter^2 inclusive will be allowed.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit [MlU]/milliliter [mL] and estradiol <40 picogram [pg]/mL [<147 picomoles /litre] is confirmatory]..
* Male subjects with female partners of child-bearing potential must agree to use contraception method. This criterion must be followed from the time of the first dose of study medication until the follow up visit.his criterion must be followed from the time of the first dose of study medication until the follow up visit (7 to 14 days post last dose).
* Aspartate Amino Transferase (AST), Alanine Amino Transferase (ALT), alkaline phosphatase, bilirubin, and creatinine less than the upper limits of normal. TSH within normal reference range. At the discretion of the principle investigator (PI) or sub-PI, these values may be repeated once.
* White blood cell count (including neutrophil counts), hemoglobin, platelets and reticulocytes greater than the lower limits of normal. At the discretion of the PI or sub-PI, these values may be repeated once.
* The subject's systolic blood pressure is inside the range of 90-140 millimeters of mercury (mmHg,) and diastolic blood pressure is inside the range of 45-90 mmHg. Heart rate is inside the range of 50-100 beat per minute (bpm) for female subjects or 45-100 bpm for male subjects.

Exclusion Criteria:

* Subject is mentally or legally incapacitated.
* Family history of prolonged QT syndrome (Torsade de Pointes) or sudden cardiac death; first-degree relative with myocardial infarction at premature age (<45 years for male relative; <55 years for female relative).
* History of or active diagnosis of diabetes mellitus.
* History of or active diagnosis of thyroid disease.
* History of or active diagnosis of pulmonary disease such as asthma, emphysema, chronic obstructive pulmonary disease or interstitial lung disease.
* History of regular alcohol consumption within 6 months of the study defined as:

Australian standard: An average weekly intake of >21 units for males and >14 units for females. One unit is equivalent to 10 g of alcohol: 270mL of full strength beer (4.8%), 375mL of mid strength beer (3.5%),470mL of light beer (2.7%), 250mL pre-mix full strength spirit (5%), 100mL of wine (13.5%) and 30mL of spirit (40%).

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* A positive Hepatitis C antibody
* A positive pre-study Hepatitis B surface antigen.
* A positive test for HIV antibody
* History of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit or indication of tobacco use as evidenced by a positive urine cotinine test at screening.
* A positive pre-study drug/alcohol screen. Unwilling to refrain from use of the illicit drugs and adhere to other protocol-stated restrictions while participating in the study. Pregnant females as determined by positive urine or serum human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* QT interval corrected for heart rate (Fridericia's)> 450 milliseconds (msec); or QTc >480 msec in subjects with Bundle Branch Block.
* Holter monitoring shows one or more of the following:
* Any symptomatic arrhythmia (except isolated extra systoles).
* Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, Supraventricular tachycardia (SVT) (>10 consecutive beats).
* Sinus tachycardia (or supraventricular tachycardia) greater than 150 bpm
* Non-sustained or sustained ventricular tachycardia (defined as >3 consecutive ventricular ectopic beats).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, Atrioventicular (AV) block [2nd degree or higher in an awake subject], Wolff-Parkinson-White (WPW) syndrome, other pre-excitation syndromes).
* Symptomatic sinus pause or sinus pause >3 seconds - unless patient is straining, vomiting, or having some other type of hypervagal response.
* 300 or more supraventricular ectopic beats in 24 hours.
* 250 or more ventricular ectopic beats in 24 hours
* Ischemia, diagnosed by a sequence of ECG changes that include flat or down sloping ST-segment depression >0.1 millivolts (mV), with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule).
* Unable to use spirometry equipment correctly.
* Abnormal spirometry results: Volume that has been exhaled at the end of the first second of forced expiration (FEV1 ) less than 80% of predicted value, FEV1/ Forced Vital Capacity: the determination of the vital capacity from a maximally forced expiratory effort (FVC )less than 70%
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 5 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the collection of adverse events (AEs). | Screening to 7-14 days post last-dose
  AEs will be collected from the start of Study Treatment and until 7-14 days post last-dose (at follow up).
Safety as assessed by hematology, clinical chemistry, urinalysis, vital signs, electrocardiogram (ECG) intervals, ECG rhythm telemetry, pulmonary function tests, respiratory rate and lung auscultation. | Pre-dose to 7-14 days post last-dose
  Absolute values and changes over time of hematology, clinical chemistry, urinalysis, vital signs (blood pressure [BP], FSH/Estradiol (Women), Urine β-hCG (Women) temperature, and heart rate), 12 LED ECG, and Holter monitoring, ECG intervals, ECG rhythm, and telemetry will be measured. Telemetry is the continuous monitoring of a subject's heart rate and rhythm from a remote location. Pulmonary function testing includes a group of tests that measure how well the lung is functioning.

SECONDARY OUTCOMES:
Composite of pharmacokinetics (PK) parameters following single dose administration of GSK2878175. | Part 1 and Day 1for Part 2
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinity]), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC [0-t]), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), observed concentration at 24hour post-dose (C24), lag time before observation of drug concentrations in sampled matrix (tlag), terminal half-life (t1/2), apparent oral clearance (CL/F).
Composite of PK parameters following repeat dose administration of GSK2878175. | on Part 2 Day 7
  PK parameters include: AUC (0-infinity), AUC (0-t), Cmax, and Ctau (Pre-dose trough concentration at the end of the dosing interval),tmax, tlag, t1/2, CL/F
Dose proportionality of GSK2878175 PK parameters following single and repeat administration | Pre-dose, Day1 and Day 7
  GSK2878175 PK parameters: AUC (0-infinity), AUC (0-t), Cmax, and Ctau (Pre-dose trough concentration at the end of the dosing interval),tmax, tlag, t1/2
The effect of a moderate fat/caloric meal on the relative bioavailability of a given single dose of GSK2878175 | Pre-dose, Day1
  GSK2878175 PK parameters: AUC (0-infinity), AUC (0-t), Cmax, and Ctau (Pre-dose trough concentration at the end of the dosing interval), tmax, tlag, t1/2, with and without moderate fat/calorie meal (Part 1).
Estimate GSK2878175 accumulation and time invariance | Pre-dose, Day1 and Day 7
  GSK2878175 AUC(0 t), Cmax, and Ctau on the last day of dosing compared to AUC(0-24), Cmax, and C24 on Day 1 to estimate accumulation ratio (R) and GSK2878175 AUC(0 t) on the last day of dosing compared to AUC(0 infinity) on Day 1 to evaluate time invariance (Part 2)
To assess attainment of steady state following repeat administration | Pre-dose, Day 1 and Day 7
  Pre-dose concentrations on Day 3 through 7 and Ctau on Day 7 to assess the achievement of steady state of GSK2878175 following repeat administration (Part 2).
To describe exposure-response relationships for various safety parameters, if appropriate. | Pre-dose, Day1 and Day 7
  Correlation between PK parameters and various safety parameters, if appropriate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 116973 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116973?search=study&search_terms=116973#rs